CLINICAL TRIAL: NCT03038815
Title: The Influence of Stability Boots on Gait Pattern in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Biomechanics, ETH Zürich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Stability Boots
Record Dates: First submitted 2017-01-25; First posted 2017-02-01 (Estimated); Results first posted 2019-11-01 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Rehabilitation After Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Controll-VACOped-Ortho Tri (Experimental): All participants are in the control and the two intervention group. The instant change of the ankle joint motion is analyzed. For control, the participants are wearing Sport shoes.This group had the VACOped as the first intervention.
  Interventions: Device: VACOped; Device: Ortho Tri
- Controll-Ortho Tri-VACOped (Experimental): All participants are in the control and the two intervention group. The instant change of the ankle joint motion is analyzed. For control, the participants are wearing Sport shoes.This group had the Ortho Tri first intervention
  Interventions: Device: VACOped; Device: Ortho Tri

INTERVENTIONS:
Device: VACOped — restriction of ankle joint motion
Device: Ortho Tri — restriction of ankle joint motion

SUMMARY:
After an ankle injury like distorsions, fractures or arthrodeses, or congenital defects ankle support limit the range of motion in the joint, help pain relief, control loading of the injured tissues and promote recovery of a normal gait pattern. Gait analysis is applied in orthopedics, sport science and rehabilitation. Numerous measure systems and methods enable accurate analysis of human movement.

The study is set to describe and compare the gait analysis of two modifiable stability boots (Ortho® Tri-Phase and the VACOped®) on the standard walking parameters during two conditions (level and ramp walking) in healthy adults and draw comparisons with a control indoor shoe.

DETAILED DESCRIPTION:
The participants are joining one session in the gait lab. Here the are measured during walking with normal shoes and two modifiable stability boots. The duration of a session is typically 3 hours.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* 18-45 years old
* shoe size 5,6,9 or 10

Exclusion Criteria:

* injuries of the lower limbs
* previous surgeries on the lower limbs
* neuromuscular disorders
* restriction in gait capabilities
* current medical treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvio Lorenzetti, PhD, Principal Investigator — Institute for Biomechanics
Locations (1):
- Institute for Biomechanics ETH Zürich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Controll-VACOped-Ortho Tri: VACOped first
- Controll-Ortho Tri-VACOped: Ortho Tri first
Period: Controll Condition, 1 Hour
Arm/Group | Controll-VACOped-Ortho Tri | Controll-Ortho Tri-VACOped
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Intervention 1, 1 Hour
Arm/Group | Controll-VACOped-Ortho Tri | Controll-Ortho Tri-VACOped
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0
Period: Intervention 2, 1 Hour
Arm/Group | Controll-VACOped-Ortho Tri | Controll-Ortho Tri-VACOped
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Group-VACOped-Ortho Tri-Phase: All participants are in the control and the two intervention group. The instant change of the ankle joint motion is analyzed. For control, the participants are wearing Sport shoes.
  This group had the VACUped as first intervention.
- Control Group-Ortho Tri-Phase-VACOped: All participants are in the control and the two intervention group. The instant change of the ankle joint motion is analyzed. For control, the participants are wearing Sport shoes.
  This group had the Ortho Tri as first intervention.
- Total: Total of all reporting groups
Arm/Group | Control Group-VACOped-Ortho Tri-Phase | Control Group-Ortho Tri-Phase-VACOped | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24 (2) | 24 (2) | 24 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 5 | 5 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: ROM Ankle Joint
Description: Ankle joint motion ROM Sagittal left, during gait
Time Frame: duration of a session is typically 3 hours
Measure: Mean (Standard Deviation); unit: degree
Groups:
- Control Group: All participants are in the control and the two intervention group. The instant change of the ankle joint motion is analyzed. For control, the participants are wearing Sport shoes.
- VACOped: All participants are in the control and the two intervention group. The instant change of the ankle joint motion is analyzed.
  VACOped: restriction of ankle joint motion
- Ortho Tri-Phase: All participants are in the control and the two intervention group. The instant change of the ankle joint motion is analyzed.
  Ortho Tri-Phase: restriction of ankle joint motion
Arm/Group | Control Group | VACOped | Ortho Tri-Phase
Number analyzed (Participants) | 20 | 20 | 20
degree | 31.4 (5.7) | 18.4 (3.5) | 21.2 (3.7)

2. Secondary Outcome: Symmetrie Index
Description: The symmetrie index, represents the % difference step length, index= 2*100*(step length left-step length right)/(step length left+step length right) This measure has no unit. 0 would represent a total symmetric gait.
Time Frame: duration of a session is typically 3 hours
Measure: Mean (Standard Deviation); unit: percentage of step length
Arm/Group | Control Group | VACOped | Ortho Tri-Phase
Number analyzed (Participants) | 20 | 20 | 20
percentage of step length | 2.45 (0.05) | 7.62 (0.15) | 1.9 (0.04)

ADVERSE EVENTS:
Time Frame: during the intervention, up to 3 hours
Description: Standard definitions
Groups:
- Controll-VACOped-Ortho Tri: This group had first the control condition, than the VACUped intervention and last the Ortho Tri intervention.
- Controll-Ortho Tri-VACOped: This group had first the control condition, than the Ortho Tri intervention and last the VACOped intervention.
Arm/Group | Controll-VACOped-Ortho Tri | Controll-Ortho Tri-VACOped
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT03038815/Prot_SAP_000.pdf